CLINICAL TRIAL: NCT04208997
Title: Continuation of Antiarrhythmics Following caThEteR Ablation for Ventricular Tachycardia (AFTER-VT) Trial: A Pilot Randomized Clinical Trial
Brief Title: Continuation of Antiarrhythmics Following Ventricular Tachycardia Catheter Ablation
Acronym: AFTER-VT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated due to low accrual
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Arvindh Kanagasundram, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 191113
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Results first posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Tachycardia, Ventricular; Catheter Ablation
Keywords: Ventricular Tachycardia; Catheter Ablation; Antiarrhythmic drugs
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Anti-Arrhythmia Agents; Amiodarone; Sotalol

STUDY DESIGN:
Intervention Model Description: Patients that meet inclusion criteria and agree to participate will be randomized and allocated to continue class III AADs or discontinuation using block randomization, stratified by type of AADs and type of cardiomyopathy (ischemic vs nonischemic) used until goal enrollment is achieved. The randomization sequence was created using STATA 14.2 (StataCorp, College Station, TX, USA) statistical software.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuation of antiarrhythmic drugs (Experimental): Patients will continue the class III antiarrhythmic drug they were receiving prior the VT catheter ablation for 3 months after the ablation.
  Interventions: Drug: Antiarrhythmic drug
- Discontinuation of antiarrhythmic drugs (No Intervention): Patients will stop class III antiarrhythmic drug they were receiving prior to the VT catheter ablation.

INTERVENTIONS:
Drug: Antiarrhythmic drug — Continuation of amiodarone or sotalol.
  Other Names: Amiodarone; Sotalol
  Arms: Continuation of antiarrhythmic drugs

SUMMARY:
The investigators aim to study if patients that undergo catheter ablation for ventricular tachycardia benefit from continuation of Vaughan-Williams class III antiarrhythmic drugs for 3 months after their ablation.

DETAILED DESCRIPTION:
Catheter ablation is a valuable option to control recurrent Ventricular Tachycardia (VT) in patients with structural heart disease. A recent trial proved that catheter ablation is superior to escalation of anti arrhythmic drugs (AADs) in prevention of VT recurrence and death (Sapp et al. N Engl J Med 2016; 375:111-121). However, even with ablation, approximately 20-50% of patients will have an episode of VT within one year. This is probably explained in part by the substrate (myocardial scar from cardiomyopathy) persists after VT ablation and that ablation lesions heal and evolve over days, weeks and even months. Most patients (if not all) of patients who undergo ablation are on AADs and usually have failed at least one of them. Furthermore, most AADs, and Vaughan Williams class III AADs in particular (the most frequently used to treat VT) carry significant and life-threatening side effects from pulmonary, hepatic and hematologic toxicities up to significant ventricular arrhythmias and death. Since these patients have already failed AADs, and the significant adverse profile of AADs, there is no evidence that the benefits of continuation of these drugs will surpass the risks after ablation. Therefore the investigators decided to ask the question:

Among patients with structural heart disease who undergo VT ablation, does continuation of class III AADs for 3 months, increases VT-free survival compared to discontinuation of antiarrhythmic drug therapy?

Based on expert consensus about clinical equipoise in regards of AAD continuation after VT ablation, the investigators decided to select patients with lowest risk of VT recurrence after ablation as our study population. The investigators aim to include in our study only those patients who have an Implantable Cardioverter-Defibrillator (ICD), who have NO inducible VT at the end of the ablation procedure and also who have NO inducible VT prior to discharge on a procedure called non-invasive programmed stimulation (NIPS). It has been shown that patients with inducible VT at the end of ablation and during NIPS have significantly higher risk of VT recurrence compared to those in whom VT was not induced. In NIPS, one uses the previously Implanted ICD to pace the ventricle fast enough to try to induce VT. Both procedures will be performed as usual practice in patients who undergo VT ablation in the arrhythmia service.

The specific aim of this pilot study is to evaluate whether the strategy of continuation of class III AADs following initial catheter ablation for VT, improves VT-free survival and reduces readmissions.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years.
2. Able to give written, informed consent
3. Structural heart disease.
4. Implanted and normally functioning ICD or undergoing ICD implant at index admission.
5. Undergoing initial radiofrequency ablation procedure for sustained monomorphic VT.
6. Receiving a class III AADs prior to VT ablation.
7. No VT inducible at the end of VT ablation.
8. No VT inducible on non-invasive programmed stimulation following VT ablation.

Exclusion Criteria:

1. LV assist device in place
2. Decompensated heart failure and/or requiring continuous inotropic therapy and/or awaiting cardiac transplantation
3. Ongoing acute coronary syndrome.
4. Mechanical prosthetic aortic and mitral valves.
5. Pedunculated or mobile left ventricular thrombus.
6. Persistent VT at the end of index catheter ablation.
7. Absolute contraindications for class III AADs.
8. Participation in other trial.
9. VT induced on NIPS after VT ablation.
10. Another reason for continuation of class III AADs (i.e., atrial fibrillation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arvindh Kanagasundram, M.D, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Continuation of Antiarrhythmic Drugs | Discontinuation of Antiarrhythmic Drugs
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuation of Antiarrhythmic Drugs | Discontinuation of Antiarrhythmic Drugs | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61.2 [58.3 to 62.6] | 69.1 [66.8 to 71.5] | 64 [61.2 to 64.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5
Cardiomyopathy type [Count of Participants; unit: Participants]
  Ischemic cardiomyopathy | 3 | 2 | 5
  Dilated cardiomyopathy | 0 | 0 | 0
Left Ventricular Ejection Fraction (LVEF) [Median (Inter-Quartile Range); unit: %] | 25 [25 to 32.5] | 42.5 [36.3 to 48.8] | 30 [25 to 40]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Dead or With VT Recurrence at One Year
Description: A composite of all-cause mortality and VT recurrence one year after index VT ablation
Time Frame: One year after ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Continuation of Antiarrhythmic Drugs | Discontinuation of Antiarrhythmic Drugs
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

2. Secondary Outcome: All-cause Mortality
Description: Deaths by any cause one year after ablation
Time Frame: One year after ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Continuation of Antiarrhythmic Drugs | Discontinuation of Antiarrhythmic Drugs
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

3. Secondary Outcome: Number of Participants With VT Recurrence
Description: Self-terminating sustained VTs (>30 seconds or hemodynamic instability) and VT requiring ICD device therapies for termination (appropriate therapies) will be considered VT recurrences
Time Frame: One year after ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Continuation of Antiarrhythmic Drugs | Discontinuation of Antiarrhythmic Drugs
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With VT/Electrical Storm
Description: Three or more episodes of sustained VT, ventricular fibrillation, or appropriate ICD therapies within a 24-hour period
Time Frame: One year after ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Continuation of Antiarrhythmic Drugs | Discontinuation of Antiarrhythmic Drugs
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With Readmission for Heart Failure
Description: Admissions with heart failure as principal diagnosis
Time Frame: One year after ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Continuation of Antiarrhythmic Drugs | Discontinuation of Antiarrhythmic Drugs
Number analyzed (Participants) | 3 | 1
Participants | 0 | 0

6. Other Pre Specified Outcome: Number of Participants With Drug Side Effects
Description: Side effects attributed to any drug of the patient's regimen
Time Frame: One year after ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Continuation of Antiarrhythmic Drugs | Discontinuation of Antiarrhythmic Drugs
Number analyzed (Participants) | 3 | 2
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Chart review
Arm/Group | Continuation of Antiarrhythmic Drugs | Discontinuation of Antiarrhythmic Drugs
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 1/3 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuation of Antiarrhythmic Drugs (N=3) | Discontinuation of Antiarrhythmic Drugs (N=2)
Fatigue (Nervous system disorders) | 1 (1) | 0 (0) — Fatigue and asthenia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT04208997/Prot_SAP_001.pdf